CLINICAL TRIAL: NCT03780127
Title: ZX008 Expanded Access Protocol - Dravet Syndrome Treatment Plan
Brief Title: ZX008 Expanded Access Protocol
Status: Approved for marketing | Type: Expanded Access
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: ZX008-1800
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Fenfluramine

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Fenfluramine Hydrochloride — ZX008 drug product is an oral aqueous solution of fenfluramine hydrochloride. The product is sugar free and is intended to be compatible with KD.
  Other Names: ZX008

SUMMARY:
The treatment plan for this Expanded Access Protocol is for patients with Dravet syndrome who do not qualify for participation in one of the ongoing ZX008 clinical trials.

DETAILED DESCRIPTION:
The treatment plan consists of an up to 24-month Treatment Period. Access is via application by your health care provider and available at one of the Expanded Access treatment centers. The dose of ZX008 for the duration of the Treatment Period will range from 0.2 mg/kg/day to a maximum of 0.8 mg/kg/day, not to exceed a total daily dose of 30 mg/day; for patients concurrently being prescribed stiripentol, the maximum will be 0.5mg/kg/day, not to exceed a total daily dose of 20 mg/day.

The fenfluramine US Expanded Access Program (US EAP) is available to full-time US Residents only.

Participation in the US EAP is limited to patients currently residing in the US. Residency in the US must be for the duration of participation in the US EAP. Drug may not be shipped outside the US.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, age 2 years and older, inclusive as of Study Day 1.
* Patient is diagnosed with Dravet syndrome.
* Patient is experiencing convulsive seizures which are not controlled by current AEDs.
* Patient is receiving at least one AED and will remain on at least one AED for the duration of treatment.
* Patient has been approved for inclusion by Zogenix.

Exclusion Criteria:

* Patient requires or starts using an unacceptable or contraindicated concomitant medication.
* Patient has valvulopathy.
* Patient is at risk for pulmonary hypertension.
* Patient exclusion will be at the sole discretion of the Sponsor.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Derived] Cross JH, Galer BS, Gil-Nagel A, Devinsky O, Ceulemans B, Lagae L, Schoonjans AS, Donner E, Wirrell E, Kothare S, Agarwal A, Lock M, Gammaitoni AR. Impact of fenfluramine on the expected SUDEP mortality rates in patients with Dravet syndrome. Seizure. 2021 Dec;93:154-159. doi: 10.1016/j.seizure.2021.10.024. Epub 2021 Nov 2. PMID 34768178